CLINICAL TRIAL: NCT02901925
Title: A Phase 0 Open Label, Single-center Clinical Trial of ABY-029, an Anti-EGFR Fluorescence Imaging Agent Via Single Intravenous Injection to Subjects With Recurrent Glioma
Brief Title: A Microdose Evaluation Study of ABY-029 in Recurrent Glioma
Acronym: ABY-029
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Dartmouth College (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David W. Roberts, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D16107; R01CA167413 (NIH)
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Results first posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-08

CONDITIONS: Glioma
Keywords: ABY-029; Affibody; Molecular Fluorescence-Guided Surgery; Epidermal Growth Factor Receptor (EGFR)
MeSH Terms: conditions — Glioma | interventions — ABY-029

STUDY DESIGN:
Intervention Model Description: Pilot feasibility study
Masking Description: open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ABY-029 1X dose group (Experimental): ABY-029 will be administered at the 1X dose level prior to surgery. Probe will be used in vivo to determine if signal is detectable, and ex vivo tissue pathology will measure extent of binding with EGFR positive tumor tissue.
  Interventions: Drug: ABY-029
- ABY-029 3X dose group (Experimental): ABY-029 will be administered at the 3X dose level prior to surgery. Probe will be used in vivo to determine if signal is detectable, and ex vivo tissue pathology will measure extent of binding with EGFR positive tumor tissue.
  Interventions: Drug: ABY-029
- ABY-029 6X dose group (Experimental): ABY-029 will be administered at the 6X dose level prior to surgery. Probe will be used in vivo to determine if signal is detectable, and ex vivo tissue pathology will measure extent of binding with EGFR positive tumor tissue.
  Interventions: Drug: ABY-029

INTERVENTIONS:
Drug: ABY-029 — Using a sample size of 6-12 patients, ABY-029 will be administered via single intravenous injection to subjects with recurrent glioma, approximately 1-3 hours prior to surgery. Microdose levels of ABY-029 have been selected to determine if a fluorescence signal can be detected by wide-field imaging technology with a signal-to-noise ratio of 10, which is considered necessary for subsequent assessment of diagnostic performance of ABY-029 as a tumor biomarker sufficient to guide surgical resection in the future. Administration of the study drug is not intended to alter the extent of planned brain tumor resection during the surgical procedure.
  Other Names: ABY-029 trifluoroacetate salt; IRDye® 800CW Maleimide labeled Affibody peptide

SUMMARY:
The primary study objective is to determine if microdoses of ABY-029 lead to detectable signals in sampled tissues with an EGFR pathology score ≥ 1 based on histological staining.

The secondary study objective is to assess diagnostic accuracy of ABY-029 detection by iFI and intraoperative probe relative to histopathology diagnosis, and other indicators (e.g. proliferation, infiltration, etc.) as the gold standard, and to measure the molecular uptake and concentration of ABY-029 in resected specimens.

DETAILED DESCRIPTION:
The investigators plan a sample size of 6-12 patients in this open label, single center, clinical trial of ABY-029. Administration will occur as a single intravenous injection to subjects with recurrent glioma, approximately 1-3 hours prior to surgery.

The protocol is not a safety study since no physiological effects are expected at microdose levels of ABY-029. Rather, doses have been selected to determine if a fluorescence signal can be detected by wide-field imaging technology with a signal-to-noise ratio of 10, which is considered necessary for subsequent assessment of diagnostic performance of ABY-029 as a tumor biomarker sufficient to guide surgical resection in the future. No diagnostic or therapeutic intent is proposed, and administration of the study drug is not intended to alter the extent of planned brain tumor resection during the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative diagnosis of recurrent high-grade glioma having EGFR positive tissue from prior surgery.
2. Tumor judged to be suitable for open cranial resection based on preoperative imaging studies.
3. Valid informed consent by subject.
4. Age ≥ 18 years old.

Exclusion Criteria:

1. Pregnant women or women who are breast feeding.
2. Patients on any experimental anti-EGFR targeted therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David W Roberts, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited and enrolled at 1 academic medical center between February 2017 and June 2021. Of 14 participants enrolled (patients met the inclusion criteria and signed the consent form), a total of 12 received the study drug and started the study across the 3 dose groups: 3 patients in the 1X dose group, 3 patients in the 3X dose group, and 6 patients in the 6X dose group.
Groups:
- ABY-029 1X Dose Group: A 1X dose of ABY-029 will be administered prior to surgery. Probe will be used in vivo to determine if signal is detectable, and ex vivo tissue pathology will measure extent of binding with EGFR positive tumor tissue.
  ABY-029: In 3 patients, ABY-029 will be administered via single intravenous injection to subjects with recurrent glioma, approximately 1-3 hours prior to surgery. Microdose levels of ABY-029 have been selected to determine if a fluorescence signal can be detected by wide-field imaging technology with a signal-to-noise ratio of 10, which is considered necessary for subsequent assessment of diagnostic performance of ABY-029 as a tumor biomarker sufficient to guide surgical resection in the future. Administration of the study drug is not intended to alter the extent of planned brain tumor resection during the surgical procedure.
- ABY-029 3X Dose Group: A 3X dose of ABY-029 will be administered prior to surgery. Probe will be used in vivo to determine if signal is detectable, and ex vivo tissue pathology will measure extent of binding with EGFR positive tumor tissue.
  ABY-029: In 3 patients, ABY-029 will be administered via single intravenous injection to subjects with recurrent glioma, approximately 1-3 hours prior to surgery. Microdose levels of ABY-029 have been selected to determine if a fluorescence signal can be detected by wide-field imaging technology with a signal-to-noise ratio of 10, which is considered necessary for subsequent assessment of diagnostic performance of ABY-029 as a tumor biomarker sufficient to guide surgical resection in the future. Administration of the study drug is not intended to alter the extent of planned brain tumor resection during the surgical procedure.
- ABY-029 6X Dose Group: A 6X dose of ABY-029 will be administered prior to surgery. Probe will be used in vivo to determine if signal is detectable, and ex vivo tissue pathology will measure extent of binding with EGFR positive tumor tissue.
  ABY-029: In 3-6 patients, ABY-029 will be administered via single intravenous injection to subjects with recurrent glioma, approximately 1-3 hours prior to surgery. Microdose levels of ABY-029 have been selected to determine if a fluorescence signal can be detected by wide-field imaging technology with a signal-to-noise ratio of 10, which is considered necessary for subsequent assessment of diagnostic performance of ABY-029 as a tumor biomarker sufficient to guide surgical resection in the future. Administration of the study drug is not intended to alter the extent of planned brain tumor resection during the surgical procedure.
Period: Overall Study
Arm/Group | ABY-029 1X Dose Group | ABY-029 3X Dose Group | ABY-029 6X Dose Group
Started | 3 | 3 | 6
Completed | 3 | 3 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ABY-029 1X Dose Group: A 1X dose of ABY-029 will be administered prior to surgery. Probe will be used in vivo to determine if signal is detectable, and ex vivo tissue pathology will measure extent of binding with EGFR positive tumor tissue.
  ABY-029: Using a sample size of 3 patients, ABY-029 will be administered via single intravenous injection to subjects with recurrent glioma, approximately 1-3 hours prior to surgery. Microdose levels of ABY-029 have been selected to determine if a fluorescence signal can be detected by wide-field imaging technology with a signal-to-noise ratio of 10, which is considered necessary for subsequent assessment of diagnostic performance of ABY-029 as a tumor biomarker sufficient to guide surgical resection in the future. Administration of the study drug is not intended to alter the extent of planned brain tumor resection during the surgical procedure.
- ABY-029 3X Dose Group: A 3X dose of ABY-029 will be administered prior to surgery. Probe will be used in vivo to determine if signal is detectable, and ex vivo tissue pathology will measure extent of binding with EGFR positive tumor tissue.
  ABY-029: Using a sample size of 3 patients, ABY-029 will be administered via single intravenous injection to subjects with recurrent glioma, approximately 1-3 hours prior to surgery. Microdose levels of ABY-029 have been selected to determine if a fluorescence signal can be detected by wide-field imaging technology with a signal-to-noise ratio of 10, which is considered necessary for subsequent assessment of diagnostic performance of ABY-029 as a tumor biomarker sufficient to guide surgical resection in the future. Administration of the study drug is not intended to alter the extent of planned brain tumor resection during the surgical procedure.
- ABY-029 6X Dose Group: A 6X dose of ABY-029 will be administered prior to surgery. Probe will be used in vivo to determine if signal is detectable, and ex vivo tissue pathology will measure extent of binding with EGFR positive tumor tissue.
  ABY-029: Using a sample size of 3-6 patients, ABY-029 will be administered via single intravenous injection to subjects with recurrent glioma, approximately 1-3 hours prior to surgery. Microdose levels of ABY-029 have been selected to determine if a fluorescence signal can be detected by wide-field imaging technology with a signal-to-noise ratio of 10, which is considered necessary for subsequent assessment of diagnostic performance of ABY-029 as a tumor biomarker sufficient to guide surgical resection in the future. Administration of the study drug is not intended to alter the extent of planned brain tumor resection during the surgical procedure.
- Total: Total of all reporting groups
Arm/Group | ABY-029 1X Dose Group | ABY-029 3X Dose Group | ABY-029 6X Dose Group | Total
Number analyzed (Participants) | 3 | 3 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 3 | 7
  >=65 years | 2 | 0 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 4 | 6
  Male | 1 | 3 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 2 | 6 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Fluorescence Signal Detection
Description: The primary study endpoint is to determine if the fluorescence signal from ABY-029, as measured by Biological Variance Ratio (BVR), can be detected in brain tissue during surgery. This will help researchers determine if ABY-029 functions well for imaging brain tumor tissue during surgery.
Time Frame: during procedure
Measure: Mean (Standard Deviation); unit: Biological variance ratio
Groups:
- 1X Dose Group: Patients received 30 nanomoles or 237µg of ABY-029
- 3X Dose Group: Patients received 90 nanomoles or 711µg of ABY-029
- 6X Dose Group: Patients received 180 nanomoles or 1.42 mg of ABY-029
Arm/Group | 1X Dose Group | 3X Dose Group | 6X Dose Group
Number analyzed (Participants) | 3 | 3 | 6
Biological variance ratio | 6.2 (2.4) | 5.0 (1.2) | 8.8 (3.7)

2. Secondary Outcome: Mean Tumor-to-background Ratio
Description: A secondary study endpoint is to calculate the ratio of the average (mean) fluorescence intensity of ABY-029 measured in the tumor, to the average (mean) fluorescence intensity of ABY-029 measured in the surrounding tissues in the brain during surgery. This will help researchers determine how well ABY-029 works for imaging tumor tissue.
Time Frame: during procedure
Measure: Mean (Standard Deviation); unit: tumor-to-background ratio
Arm/Group | 1X Dose Group | 3X Dose Group | 6X Dose Group
Number analyzed (Participants) | 3 | 3 | 6
tumor-to-background ratio | 1.7 (0.1) | 2.1 (0.6) | 2.6 (0.7)

3. Secondary Outcome: Ex Vivo Fluorescence Intensity
Description: Another secondary study endpoint is to quantify the relationship between the dose of ABY-029 administered and the fluorescence intensity produced by ABY-029 in ex vivo tissue samples after they have been transferred to the pathology department. This endpoint will be measured in relative fluorescence units, and will help researchers conduct analyses on how well ABY-029 works for imaging in tissue following surgery.
Time Frame: post surgical
Measure: Mean (Standard Deviation); unit: relative fluorescence units
Arm/Group | 1X Dose Group | 3X Dose Group | 6X Dose Group
Number analyzed (Participants) | 3 | 3 | 6
relative fluorescence units | 61.4 (25.1) | 215.2 (109.1) | 884.1 (475.4)

ADVERSE EVENTS:
Time Frame: 1 month
Groups:
- ABY-029 6X Dose Group: A 6X dose of ABY-029 will be administered prior to surgery. Probe will be used in vivo to determine if signal is detectable, and ex vivo tissue pathology will measure extent of binding with EGFR positive tumor tissue.
  ABY-029: Using a sample size of 6 patients, ABY-029 will be administered via single intravenous injection to subjects with recurrent glioma, approximately 1-3 hours prior to surgery. Microdose levels of ABY-029 have been selected to determine if a fluorescence signal can be detected by wide-field imaging technology with a signal-to-noise ratio of 10, which is considered necessary for subsequent assessment of diagnostic performance of ABY-029 as a tumor biomarker sufficient to guide surgical resection in the future. Administration of the study drug is not intended to alter the extent of planned brain tumor resection during the surgical procedure.
Arm/Group | ABY-029 1X Dose Group | ABY-029 3X Dose Group | ABY-029 6X Dose Group
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/6
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/25/NCT02901925/Prot_SAP_001.pdf
  • Informed Consent Form (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/25/NCT02901925/ICF_000.pdf